CLINICAL TRIAL: NCT07303959
Title: Sleep Treatment for Teens
Brief Title: Sleep Treatment for Teens (RCT Phase)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Old Dominion University (Other); Children's Hospital of The King's Daughters (Other)
Responsible Party: Principal Investigator, Evan M. Kleiman, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2021001233_mod 10; R34MH123590 (NIH)
Record Dates: First submitted 2025-06-23; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Sleep Problems; Suicidal Ideation; Suicidal Behavior
MeSH Terms: conditions — Parasomnias; Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (TAU) + ecological momentary assessment (EMA) (Active Comparator): Treatment as usual plus assessments via EMA
  Interventions: Behavioral: Treatment as Usual (TAU)
- Sleepio (TM) + Treatment as usual (TAU) + EMA (Experimental): Sleepio is a mobile Digital Cognitive Behavior Therapy for Insomnia (dCBT-I) app.
  Interventions: Behavioral: Sleepio; Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Sleepio — Sleepio is a mobile Digital Cognitive Behavior Therapy for Insomnia (dCBT-I) app.
  Arms: Sleepio (TM) + Treatment as usual (TAU) + EMA
Behavioral: Treatment as Usual (TAU) — Treatment as usual as part of standard inpatient care, and any outpatient care received.

SUMMARY:
The purpose of this research study is to compare (vs. treatment as usual) a brief (6-session), empirically supported, and highly disseminable version of digital (i.e., smartphone or web-based) cognitive behavioral therapy for insomnia (dCBT-I), called SleepioTM, in suicidal adolescents with co-occurring insomnia during the high-risk post-hospitalization period. Suicide is the 2nd leading cause of death among adolescents. Sleep problems, such as insomnia symptoms-the most common sleep problem in youth-may be a particularly promising treatment target to reduce suicide risk in adolescents. The investigators propose to test the feasibility, acceptability, and effectiveness of dCBT-I in a two-site (Rutgers and Old Dominion University) pilot study trial. Adolescents, 14-18 years-old, recently hospitalized for suicide risk with co-occurring insomnia (n=80, 50% at each site), will receive either dCBT-I (six weekly, 20-minute sessions) plus post-hospitalization treatment-as-usual (TAU) or TAU alone. Adolescents will complete assessments pre-treatment, during the treatment phase including at the end of treatment, and 1-month follow-up post-treatment.

ELIGIBILITY:
Inclusion:

1. Age 14-18 years old.
2. Recent hospitalization due to suicide risk (i.e., suicide attempts, aborted/interrupted attempts, or suicide ideation with intent and/or a plan) using an abbreviated version of the semi-structured and well-validated Columbia Suicide Severity Rating Scale (C-SSRS; Posner et al., 2011). Regarding recency, adolescents will need to complete the baseline within three months (Study 1) or 45 days (Study 2) of discharge in order to capture the high-risk post-discharge period, which is up to 3 months following discharge from acute psychiatric hospitalization (Chung et al., 2017).
3. Clinically significant insomnia symptoms: SCI scores ≤16 will be used to recruit a sample with clinically significant insomnia symptoms. The ISI will also be administered to gain additional information about the nature of adolescents' sleep problems in order to confirm primary insomnia. ISI scores may also be obtained via chart review when applicable
4. Access to or willingness to use a compatible Smart Device. SleepioTM works with any internet connection (cellular or Wifi) on any iOS device running iOS 10.3 or later or on any Android device running Android OS 8.0 or later. Metricwire is compatible with all devices that SleepioTM is compatible with. If an interested adolescent does not have access to their own smart device, the research team will offer them a loaner device for the duration of the treatment/follow-up phase.

Adolescents will be excluded based on the following exclusion criteria:

1. Prior CBT-I treatment, which would indicate lack of response to a prior reasonable dose of this treatment.
2. Bipolar disorder given that certain components of CBT-I (e.g., sleep restriction) may be risky for this population.
3. Substance use disorder that is primary to insomnia which would require alternative treatment.
4. Presence of factors that may reduce participants' ability to consent or complete the study procedures (e.g., current psychosis, other-directed violence; severe cognitive impairment, non-English speaking).
5. Unwillingness to wear wrist actigraphy or complete the EMA surveys.
6. Not having a parent willing to provide permission (if participant is a minor) or to consent to their own participation (required for all adolescents). Eligibility will not be based on biological sex, gender identity, race, or ethnicity. These variables will be assessed during screening to compare those who are and are not eligible.
7. Having a sibling who has enrolled in the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity | Up to 12 weeks
  Insomnia Severity Index (same measure as baseline) assessed weekly from the beginning of treatment until the treatment is complete (or a maximum of 12 weeks to match assessment with the TAU group).
Suicidal thoughts | Up to 12 weeks
  Suicide ideation severity will be measured weekly with the Beck Suicide Ideation Scale (same measure as baseline) until the end of treatment.

SECONDARY OUTCOMES:
Sleep efficiency | Daily through study completion, up to 12 weeks
  Sleep efficiency (SE), percent of time in bed spent asleep, assessed via Actiwatch.
Sleep Onset Latency | Daily throughout the study (12 weeks)
  Sleep onset latency (SOL): how many minutes it takes to fall asleep, assessed via Actiwatch device
Daily Suicidal Thoughts | Daily through study completion, up to 12 weeks
  Daily reports of suicide ideation from EMA
Wake after sleep onset | Daily through study completion, up to 12 weeks
  Wake after sleep onset (WASO): total amount of time awake during the night, assessed via Actiwatch wearable.
Subjective sleep quality | Daily through study completion, up to 12 weeks
  Sleep quality: subjective ratings on 1=very poor to 5=very good, assessed via ecological momentary assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kleiman, Principal Investigator — Rutgers
Locations (2):
- United States (2):
  - Rutgers University Behavioral Healthcare, Piscataway, New Jersey
  - Children's Hospital of The King's Daughters, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Via NIMH data archive
Supporting Information: SAP, ICF
Time Frame: 1 year after the study ends
Access Criteria: Access to the NIMH data archive

DOCUMENTS (1):
  • Informed Consent Form: new (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT07303959/ICF_000.pdf